CLINICAL TRIAL: NCT00313950
Title: Immunogenicity and Safety of AVAXIM™ 80U-Pediatric Administered Alone or Concomitantly With TRIMOVAX™ in 12-13 Months Old Healthy Hepatitis A Seronegative Turkish Children
Brief Title: Immunogenicity and Safety of Hepatitis A Vaccine Given at the Same Time of Measles, Mumps, Rubella Combined Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HAF65
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Measles; Mumps; Rubella; Hepatitis A
Keywords: measles; rubella; mumps; hepatitis A
MeSH Terms: conditions — Measles; Mumps; Rubella; Hepatitis A | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental)
  Interventions: Biological: Inactivated Hep A vaccine; Attenuated Measles Mumps Rubella
- Group 2 (Experimental)
  Interventions: Biological: Attenuated Measles Mumps Rubella; Inactivated Hep A vaccine
- Group 3 (Experimental)
  Interventions: Biological: Inactivated Hep A vaccine; Attenuated Measles Mumps Rubella

INTERVENTIONS:
Biological: Inactivated Hep A vaccine; Attenuated Measles Mumps Rubella — 0.5 mL, intramuscular (IM) (HAV Day 0 and 168); 0.5 mL, IM (MMR Day 28)
  Other Names: AVAXIM™; TRIMOVAX™
  Arms: Group 1
Biological: Attenuated Measles Mumps Rubella; Inactivated Hep A vaccine — 0.5 mL, IM (MMR, Day 0); 0.5 mL, IM (HAV Day 28 and 168)
  Other Names: TRIMOVAX™; AVAXIM™
  Arms: Group 2
Biological: Inactivated Hep A vaccine; Attenuated Measles Mumps Rubella — 0.5 mL, IM (HAV Day 0 and 168); 0.5 mL, IM (MMR, Day 0)
  Other Names: AVAXIM™; TRIMOVAX™
  Arms: Group 3

SUMMARY:
The present study will explore the immunogenicity of AVAXIM™ 80U-Pediatric in 12-13 months Turkish children and check if the administration of the MMR trivalent vaccine on the same day but at different site will interfere on immunogenicity for the four valences Hepatitis A, Measles, Mumps, and Rubella.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-13 months on the day of inclusion
* Born at full term of pregnancy (>37 weeks) with a birth weight ≥ 2.5 kg
* Informed consent form signed by the parent(s) or other legal representative
* Able to attend all scheduled visits and to comply with all trial procedures
* Subjects having received only one or no injection of vaccine against Measles
* Subjects anti-HAV seronegative according to the results obtained at the screening visit*

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the (first) trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
* Systemic hypersensitivity to any of the vaccines components or history of a life-threatening reaction to the trial vaccines or a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion
* Blood or blood-derived products received in the past 3 months
* Any vaccination in the 4 weeks preceding the first trial vaccination
* Vaccination planned in the 4 weeks following any trial vaccination
* History of hepatitis A, Mumps, Measles and/or Rubella infection (confirmed either clinically, serologically or microbiologically)
* Previous vaccination against hepatitis A with the trial vaccine or another vaccine
* Previous vaccination against Mumps, Measles and Rubella with a Mumps, Measles and Rubella trivalent combined vaccine
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* History of seizures
* Febrile illness (axillary temperature ≥37.4°C]) on the day of inclusion

Ages: 12 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 470 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of Hepatitis A Vaccine in subjects receiving Pediatric vaccines. | Day 7 - Day 196

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (1):
- Izmir, Turkey (Türkiye)

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com